CLINICAL TRIAL: NCT00644280
Title: Evaluation of Safety and Efficacy of Ranibizumab in Glaucoma Patients Treated With Filtration Tubes"
Brief Title: Ranibizumab in Preventing Failure of Ahmed Valve Glaucoma Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LinLucentis; NIH Grant # FVF4191S
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Results first posted 2013-07-26 (Estimated); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Glaucoma
Keywords: Glaucoma,Ahmed Valve
MeSH Terms: conditions — Glaucoma | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab (Active Comparator): Ranibizumab (0.5 mg in 0.05 mL) administered intravitreally at 3 time points: 9 days before Ahmed tube insertion for open-angle glaucoma, 1 month post-surgery, and 2 months post-surgery
  Interventions: Drug: Ranibizumab
- Usual care (No Intervention): Standard of care Ahmed tube insertion for open-angle glaucoma without injections of Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — intravitreal injection of 0.5 mg ranibizumab 1 week prior to tube insertion and then monthly x 2 more injections
  Other Names: Lucentis
  Arms: Ranibizumab

SUMMARY:
To determine whether ranibizumab therapy before and after tube insertion for glaucoma surgeries can maintain the patency of the tube and prevent scar formation, and increase the chances for a successful procedure compared to observation.

DETAILED DESCRIPTION:
This is a randomized, open-label, Phase I/II study of intravitreally administered ranibizumab for the treatment of tube patency in glaucoma patients.

Thirty (30) patients with severe glaucoma requiring tubes will be randomized (2:1) to either ranibizumab or observation.

Consented, enrolled subjects assigned to the treatment group will receive open-label intravitreal injection of 0.5 mg ranibizumab 1 week prior to tube insertion and then monthly x 2 more injections Sham intravitreal injections for the observation group will NOT be performed.

Study periods:

Study start date: May 1st, 2007 (estimated) Enrollment period: 6-8 months (estimated) Follow-up period: 6 months Study end Date: December 1st, 2010 (estimated)

ELIGIBILITY:
Inclusion Criteria:

1. ability to provide written informed consent and comply with study assessment for the full duration of the study.
2. age ≥ 21
3. diagnosis of glaucoma and determined to be candidate for therapy with tube insertion.

Exclusion Criteria:

1. pregnant or lactating females
2. Persons on oral contraceptives and women of child-bearing age
3. prior enrollment in the study
4. any conditions the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
5. participation in another simultaneous medical investigation or trial
6. history of active inflammatory, infectious, or idiopathic keratitis precluding view of anterior segment structures
7. previous injections of ranibizumab in either eye.
8. Persons on Plavix (clopidogrel bisulfate) and coumadin
9. Persons with uncontrolled high blood pressure
10. Persons with renal or liver disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bhisitkul, M.D., Ph.D., Study Chair — University of California, San Francisco; Rajen U Desai, Study Chair — Stanford University; Patricia Tam, Study Director — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Desai RU, Singh K, Lin SC. Intravitreal ranibizumab as an adjunct for Ahmed valve surgery in open-angle glaucoma: a pilot study. Clin Exp Ophthalmol. 2013 Mar;41(2):155-8. doi: 10.1111/j.1442-9071.2012.02836.x. Epub 2012 Sep 4. PMID 22712537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the University of California, San Francisco (UCSF) Glaucoma Service
Period: Overall Study
Arm/Group | Ranibizumab | Usual Care
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab | Usual Care | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Tube Success at 6 Months
Description: Criteria for success at 6 months postoperatively was intraocular pressure (IOP) < 18mmHg without the necessity for adjunctive medication for pressure or IOP < 15mmHg with <=1 adjunctive medication.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Ranibizumab | Usual Care
Number analyzed (Participants) | 6 | 5
percentage of participants | 83 | 40

2. Secondary Outcome: Significant Ocular Adverse Events
Description: Participants experiencing significant ocular adverse events, including endophthalmitis and rhegmatogenous retinal detachment
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Ranibizumab | Usual Care
Number analyzed (Participants) | 6 | 5
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Ranibizumab | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

LIMITATIONS AND CAVEATS:
IOP reduction may be attributable to cataract surgery instead of or in addition to ranibizumab use. Further studies, with larger sample size and longer follow-up, are needed to evaluate safety and potential efficacy of intravitreal ranibizumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes